CLINICAL TRIAL: NCT01157962
Title: Prospective, Randomized and Multicentre Study for Investigation of Valence of Sentinel Lymph Nodes Concept in Patients With Cervical Cancer ≤ 2 cm
Brief Title: Sentinel Concept in Early Stage Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Campus Mitte/ Campus Benjamin Franklin Charité university, Gynecological Oncology Ward
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EA1/207/09
Record Dates: First submitted 2010-06-22; First posted 2010-07-08 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2009-12

CONDITIONS: Cervical Cancer
Keywords: Sentinel Concept; Lymphadenectomy; Early Stage Cervical Cancer; Overall Survive; Improvement Therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Lymph Node Excision

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A Sentinel lymphadenectomy (Experimental): In group A exclusively sentinel lymphadenectomy is performed
  Interventions: Procedure: Lymphadenectomy in cervical cancer
- Group B radical pelvine lymphadenectomy (Active Comparator): in group B radical systematic pelvic lymphadenectomy is done. In patients with tumor free lymph nodes either radical hysterectomy or, in women seeking parenthood, radical trachelectomy is performed. If lymph nodes are tumor-involved systematic pelvic and paraaortic lymphadenectomy followed by primary chemoradiation is recommended.
  Interventions: Procedure: Lymphadenectomy in cervical cancer

INTERVENTIONS:
Procedure: Lymphadenectomy in cervical cancer — Sentinel lymphadenectomy vs systematic pelvic lymphadenectomy
  Other Names: Sentinel node dissection and radical pelvic dissection

SUMMARY:
Aim of present study is to inspect, if the removal alone of sentinel lymph nodes in women with early Cervix Carcinoma lead to, at equal length, overall survival like entire systematic dissection of lymph node and at the same time is accompanied with a considerably reduction of associated intra and post operative complications of lymph node dissection.

For this purpose were randomized about 1200 patients with histological assured cervix carcinoma in stages FIGO 1a1 L1 V0, FIGO 1a2 L0 or L1 V0, FIGO1b1 L0 or L1 V0= 2 cm randomization. In the branch A takes place exclusively dissection sentinel lymph node, in the branch B takes place entire pelvic lymph node dissection. Afterwards takes place in tumor free lymph nodes the removal of uterus by a radical hysterectomy or, in presence of the wish of children, radical trachelectomy. In affected tumoural lymph nodes takes place systematic pelvic and peri aortic lymph node dissection followed by primary Radiochemotherapy.

Primary end point is overall survival; this for both groups must be equal. Secondary end point is peri- and postoperative morbidity inclusive quality of life, the benefits for women must be evident with sentinel- lymph node dissection, don't have to show for both groups any significant difference.

DETAILED DESCRIPTION:
After randomization and assignment to experimental or control group lymphadenectomy is carried out.

Four different techniques can be used: 1) laparoscopic transperitoneal 2) laparoscopic retroperitoneal 3) open extraperitoneal 4) open transperitoneal. Radioactive labeling of sentinel-lymph nodes with 99technetium-marked colloid and/or patent blue is carried out. On the day prior to the operation 50mBq 99technetium or on the day of operation 10 mBq 99technetium is injected subepithelially in the cervix at 12, 3, 6 and 9 o'clock. Preoperatively 4 cc patent blue are injected in the same manner subepithelially. At the beginning of surgery parametrial tumor involvement, intrabdominal tumor dissemination, invasion of vesica-cervical and recto-vaginal septum are excluded. A lavage of cul-de-sac for cytological analysis is performed. The retroperitoneum is opened lateral of iliac vessels and blue colored lymph or radioactive nodes are removed. Sentinel- lymph node's radioactive signal is documented in counts per second (cps).

If no sentinel-lymph node is detected, complete pelvic lymph node dissection is carried out. If tumor involved pelvic lymph nodes are shown, paraaortic lymph node dissection is carried out. If sentinel- or pelvic lymph nodes are quoted as tumor free at frozen sections, radical hysterectomy or radical trachelectomy is performed. Radical hysterectomy follows in an extension a type-2 variation. In patients with positive lymph nodes in frozen section or in definitive histo-pathology primary chemoradiation is performed.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky index
* Patients aged 18-70
* Histological assured cervix cancer (Squamous epithelium- or Adenoids cancer, adenosquamous cancer)
* Stadium FIGO from 1a1 L1 V0, FIGO 1a2 L0 or L1 V0, till FIGO 1b1 L0 or L1 V0 ≤ 2cm
* Completed and signed consent form
* Cooperation qualities of patients
* Performed explanation patients and written consent

Exclusion Criteria:

* Tumour thickness > 2cm, FIGO- staging > 1b1
* Neuroendocrine tumoural or mixed types with neuroendocrine tissues
* Tumoural invasion in vascular system (V1)
* Pregnancy, during lactation women without reliable contraception during radiochemotherapy
* Existing malignant diseases (Exception: basalioma of the skin)
* Radiotherapy of pelvis in anamnesis
* Severe internal associated diseases (Myocardial infarction, Heart pathology, Heart insufficiency NYHA III/IV, Severe chronic obstructive bronchopulmonary disease, kidney insufficiency, diabetes mellitus poorly regulated, uncontrolled infections) Anaesthesia not allowed
* Psychiatric diseases, which put off participating and after care
* HIV infection, or rather AIDS disease
* Drug addicted
* Precedent motorial or sensorial Polyneuropathies>CTC grade 1

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2010-01; Primary Completion 2014-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | one year
  Primary study end point is that overall survival of patients with sentinel-concept, has not to differentiate from that one of patients with systematic lymph node dissection.

SECONDARY OUTCOMES:
morbidity | one year
  Secondary study end points are peri- und postoperative complications percentage and life quality after EORTC QLQ C-30 and local control. Local control percentage must exhibit no difference for both groups. Complications percentage and life quality must be significative better in branch with sentinel-lymph node dissection.

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University of Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Result] Altgassen C, Hertel H, Brandstadt A, Kohler C, Durst M, Schneider A; AGO Study Group. Multicenter validation study of the sentinel lymph node concept in cervical cancer: AGO Study Group. J Clin Oncol. 2008 Jun 20;26(18):2943-51. doi: 10.1200/JCO.2007.13.8933. PMID 18565880